CLINICAL TRIAL: NCT01579890
Title: A Non-blinded, Non-placebo Controlled, Compassionate Use, Open Treatment, Open-ended Program of the Safety of Pennsaid Topical Lotion (Diclofenac) in the Treatment of Osteo or Rheumatoid Arthritis
Brief Title: Compassionate Use of Pennsaid Topical Lotion (Diclofenac) in Osteo or Rheumatoid Arthritis
Status: Approved for marketing | Type: Expanded Access
Sponsor: Mallinckrodt (Industry)
Collaborators: Nuvo Research Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 105-95
Record Dates: First submitted 2012-04-16; First posted 2012-04-18 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Osteoarthritis of the Hand
MeSH Terms: interventions — Diclofenac

INTERVENTIONS:
Drug: Diclofenac — diclofenac topical lotion

SUMMARY:
This was a compassionate use, open treatment safety study of Pennsaid topical lotion (diclofenac) for osteo or rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed osteo or rheumatoid arthritis
* Oral NSAIDs were not deemed appropriate treatment
* Completed diclofenac sensitivity patch test with negative result
* Signed informed consent form

Exclusion Criteria:

* At the discretion of the physician and HPB

Sex: All
Age Groups: Child, Adult, Older Adult